CLINICAL TRIAL: NCT02718443
Title: VXM01 Phase I Pilot Study in Patients With Operable Recurrence of a Glioblastoma to Examine Safety, Tolerability, Immune and Biomarker Response to the Investigational VEGFR-2 DNA Vaccine VXM01
Brief Title: VXM01 Phase I Pilot Study in Patients With Operable Recurrence of a Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaximm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VXM01-02-DE
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VXM01 (Experimental): VXM01 10E6 or 10E7 CFU
  Interventions: Drug: VXM01

INTERVENTIONS:
Drug: VXM01 — Oral immunotherapy targeting VEGFR2

SUMMARY:
VXM01 phase I pilot study in patients with operable recurrence of a glioblastoma to examine safety, tolerability, immune and biomarker response to the investigational VEGFR-2 DNA vaccine VXM01

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, signed and dated
2. Histologically diagnosed intracranial supratentorial malignant glioma (contrast-enhancing anaplastic astrocytoma WHO Grade III or glioblastoma WHO Grade IV).
3. Male or female patients who must be post-menopausal for at least 2 years or surgically sterile.
4. Age ≥18 years
5. Evidence of tumor progression following at least one therapy regimen that must have contained radiation and chemotherapy with temozolamid, as measured by MRI
6. Candidates for a tumor reoperation
7. Neurosurgical intervention should be postponable for 30 days
8. Laboratory results (clinical chemistry, hematology, urine, liver enzymes, creatinine) without clinically relevant abnormalities
9. Patients must be able to undergo MRI
10. No concomitant medication with dexamethasone at the time of vaccination
11. No active infection at the time of vaccination
12. Karnofsky performance status >70
13. Appropriate hematologic parameters (for immunomonitoring): leukocytes ≥4.0 x 109 / L, lymphocytes ≥0.6 x 109 / L
14. Tumor samples available for pathology review, central detection of T-cell responses in the peripheral blood and in the tumor tissue
15. No medical or social conditions that may interfere with study outcome and follow-up

Exclusion Criteria:

1. Treatment in any other clinical trial within 30 days before screening
2. Known positive test results for Hepatitis B surface antigen , hepatitis C virus antibodies, human immunodeficiency virus antibodies -1/-2
3. Any other condition or treatment that, in the opinion of the investigator, might interfere with the study or current drug or substance abuse
4. Inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study
5. Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
6. Pregnancy or breast feeding
7. Positive for anti-typhoid IgG/IgM antibodies according to the onsite test on Day 0
8. Cardiovascular disease defined as:

   Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)

   Arterial thromboembolic event within 6 months before randomization including:
   * Myocardial infarction
   * Unstable angina pectoris
   * Cerebrovascular accident
   * Transient ischemic attack
9. Congestive heart failure New York Heart Association grade III to IV
10. Serious ventricular arrhythmia requiring medication
11. Clinically significant peripheral artery disease > grade 2b according to Fontaine
12. Intracranial ischemic stroke within 6 months before randomization
13. History of intracranial hemorrhage
14. Hemoptysis within 6 months before randomization
15. Esophageal varices
16. Upper or lower gastrointestinal bleeding within 6 months before inclusion (Day 0)
17. Significant traumatic injury or surgery within 4 weeks before randomization
18. Non-healing wound, incomplete wound healing, bone fracture or any history of gastrointestinal ulcers within three years before inclusion, or positive gastroscopy within 3 months before inclusion
19. Gastrointestinal fistula
20. Thrombolysis therapy within 4 weeks before randomization
21. Presence of any acute or chronic systemic infection
22. Major surgical procedures, or open biopsy within 4 weeks before randomization
23. Chronic concurrent therapy within 2 weeks before and during the treatment period up to Day 35 with:

    * Corticosteroids (except steroids for adrenal failure or emesis prophylaxis up to 4 mg daily dose) or immunosuppressive agents
    * Antibiotics
    * Bevacizumab
    * Any cancer anti-angiogenic treatment
24. Chemotherapy from screening until reoperation (Day 35)
25. Known multi-drug resistant gram-negative germ
26. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the study results or render the patient at high risk for treatment complications
27. Women of childbearing potential
28. Any condition which results in an undue risk for the patient during the study participation according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability taking into account treatment-limiting toxicities (TLTs) | 12 months
  AEs listed together with information on onset, duration, severity, seriousness, relationship to the study drug, relationship to chemotherapy and to the underlying disease, outcome, and action taken. Frequency tables by System Organ Class and preferred term.

SECONDARY OUTCOMES:
Immune Response by Enzyme Linked Immuno Spot (ELISpot) | 12 months
  Patient-individual VEGFR-2 specific T cell responses will be determined by ELISpot using cryopreserved peripheral blood mononuclear cells
Serum biomarker Response by Enzyme Linked Immuno Sorbent Assay (ELISA) | 12 months
  Biomarkers including VEGF A and Collagen IV determined from periphaeral blood samples
Vascular normalization index (VNI) including tumor perfusion acc. to Sorensen 2009 | 12 months
  Determined by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) (ktrans), dynamic susceptibility contrast imaging (DSC), blood volume maps (cerebral blood volume [CBV] of smaller vessels) and collagen IV
Tumor immune cell infiltration by tumor tissue immunohistochemistry | 35 days
  Tumor tissue immunohistochemistry staining including Evaluations of effector T cell infiltration, regulatory T-cells (Treg), myeloid derived suppressor cells (MDSC)
Tumor response or progression on MRI acc. to Response Assessment in Neuro-Oncology (RANO) criteria | 12 months
  MRI comprising the National Brain Tumor Society /EORTC protocol for gliomas
Clinical Response including time to progression, progression free survival, overall survival | 12 months
Biodistribution and shedding of VXM01 bacteria | 10 days
  Bacterial vector tissue biodistribution, persistence, and shedding of viable Ty21a bacteria (VXM01) determined by cultivation of stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, MD, Principal Investigator — Neurology Clinic and National Center for Tumor Diseases
Locations (1):
- Neurology Clinic and National Center for Tumor Diseases, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes